CLINICAL TRIAL: NCT07372131
Title: Appropriate Management of Bacteriemic Febrile Neutropenia in High-Risk Hematological Patients. Relationship Between Duration of Antibiotic Administration, Outcome and Resistance Profile
Brief Title: Antibiotic Duration and Outcomes in High-Risk Febrile Neutropenia Patients
Acronym: PERaSTrA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas University (Other)
Collaborators: Ministry of education, university and research, Italy (Unknown)
Responsible Party: Principal Investigator, Valeria Cento, Director of the Operative Unit of Microbiology and Virology, Humanitas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERaSTrA
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Bloodstream Infection; Gram Negative Infections; Bacteraemia Caused by Gram-Negative Bacteria; Febrile Neutropenia (FN)
Keywords: Antibiotics; Bloodstream Infection; Hematological patients with febrile neutropenia; Gram-negative
MeSH Terms: conditions — Sepsis; Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care antibiotic therapy with a suggested minimum duration of 10 days.
  Interventions: Other: Standard of Care Antibiotic Duration
- Personalized Duration (Experimental): Patients in this arm will receive antibiotic therapy for a duration guided by clinical stability. Antibiotics will be discontinued after 72 consecutive hours of clinical stability, defined as apyrexia (Tc < 38°C) for at least 48 hours and stable or improved qSOFA score.
  Interventions: Other: Clinical Stability-Driven Antibiotic Discontinuation Strategy

INTERVENTIONS:
Other: Clinical Stability-Driven Antibiotic Discontinuation Strategy — A therapeutic strategy where the duration of antibiotic treatment for Gram-negative bacteraemia is determined by the achievement of clinical stability (defined as apyrexia for 48h and stable/improved qSOFA score) maintained for 72 consecutive hours
  Other Names: A
  Arms: Personalized Duration
Other: Standard of Care Antibiotic Duration — This intervention follows the standard clinical practice for treating Gram-negative bacteraemia in hematological patients. The duration of therapy is not fixed by a stability-driven rule but is based on the treating physician's decision, with a suggested minimum of 10 days.
  Other Names: B
  Arms: Standard of Care

SUMMARY:
The goal of this clinical trial is to learn if a personalized duration of antibiotic therapy, based on clinical stability, is as effective as a standard duration of at least 10 days in hospitalized patients with hematologic malignancies (such as leukemia or lymphoma) who develop febrile neutropenia and Gram-negative bacteraemia.

The main questions it aims to answer are:

* Can a personalized antibiotic duration increase the number of days free from anti-Gram-negative therapy within 28 days without compromising patient safety?
* How does the duration of antibiotic therapy (short vs. prolonged) affect the rate and modality of gut microbiota reconstitution?

Researchers will compare:

* Group A (Personalized Duration): Antibiotics are stopped after the patient maintains clinical stability (no fever and stable vital signs) for 72 consecutive hours.
* Group B (Standard of Care): Antibiotics are continued for a standard duration, typically at least 10 days, based on current clinical surveys and physician decision.

Participants will:

* Be randomized to receive either the personalized or the standard duration of antibiotic therapy once a Gram-negative infection is confirmed in the blood.
* Be monitored for 28 days to assess for new fever episodes, recurrence of infection, and overall survival.
* If participating in the microbiological sub-study, provide biological samples (blood, feces, and rectal swabs) at specific time points (at the onset of fever, at the end of treatment, and at day 28).
* Undergo specialized laboratory testing (Whole Metagenomic Sequencing) on the collected samples to evaluate the evolution of their intestinal and blood microbiota and the presence of antibiotic-resistant genes.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized controlled trial. Upon confirmation of Gram-negative bacteraemia, eligible patients are randomized 1:1 to one of two treatment strategies:

* Experimental Arm (Personalized Duration): Antibiotic therapy is discontinued once the patient achieves and maintains clinical stability for 72 consecutive hours. Clinical stability is defined as apyrexia (Tc < 38°C) for at least 48 hours and a stable or improving qSOFA score.
* Control Arm (Standard of Care): Antibiotic therapy duration follows local clinical practice, with a suggested minimum duration of 10 days, consistent with current European and Asian hematological guidelines.

In parallel, a prospective observational microbiological sub-study will utilize Shotgun Metagenomic Next-Generation Sequencing (mNGS) to analyze the evolution of the intestinal and blood microbiota. The goal is to compare the rate of MDR organism colonization and the reconstitution of the healthy microbiome between the two antibiotic duration strategies.

All participants will undergo clinical monitoring until day 28. For those enrolled in the sub-study, biological samples (stool, rectal swabs, and blood) will be collected at baseline (V1), at the end of treatment (V4), and at the end of the study (V5). These samples will be analyzed to identify clinically significant bacteria and antibiotic-resistance genes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a hematologic malignancy that is candidate for treatment with chemotherapy or bone marrow transplantation or chimeric antigen receptor T cell therapy (CAR-T)
* Diagnosis of febrile neutropenia defined according to the guidelines of the Infectious Disease Society of America, IDSA; ref: Freifeld, A.G., et al., Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis, 2011. 52(4): p. e56-93.) as: Fever: single record of oral temperature >=38.3°C or a temperature >=38.0°C sustained over a period of one hour; Neutropenia: absolute neutrophil count < 1000 cells/microL; Expected duration of neutropenia >= 7 days
* Diagnosis of bacteraemia defined by positive blood cultures (at least 1 vial positive for a non-contaminating microorganism)
* Isolation of Gram-Negative species

Exclusion Criteria:

* Contextual diagnosis of pneumonia
* Contextual diagnosis of intra-abdominal infection, in particular: neutropenic enterocolitis/typhlitis or biliary tract infection
* Persistently positive blood cultures at randomization
* Any condition that endangers the safety of the patient based on the judgment of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Days Free from Anti-Gram-Negative Antibiotic Therapy within 28 days | From the date of index blood culture collection (Day 0) up to Day 28
  Number of days that the participant is alive and free from any anti-Gram-negative antibiotic therapy, calculated from the date of the index blood culture collection (onset of infection) up to Day 28. Antibiotics active exclusively on Gram-positive bacteria (e.g., glycopeptides, daptomycin) and fluoroquinolone prophylaxis are excluded from this calculation.

SECONDARY OUTCOMES:
Incidence of New Fever Episodes | From the end of antibiotic therapy up to Day 28
  Number of participants experiencing a new episode of fever (Tc ≥ 38.3°C) occurring after a period of apyrexia of at least 72 hours
28-day All-cause Mortality | Up to Day 28
  Number of participants who died from any cause within 28 days from the onset of the index infection (date of first positive blood culture)
Relapse of Bloodstream Infection (BSI) by the Same Pathogen | From the end of antibiotic therapy up to Day 28
  Number of participants with a new positive blood culture for the same Gram-negative pathogen identified in the index episode
Recurrent BSI by Gram-negative Bacteria | From the end of antibiotic therapy up to Day 28
  Number of participants experiencing a new episode of bloodstream infection caused by any Gram-negative bacteria different from the index pathogen
Emergence of Multi-Drug Resistant Organisms (MDRO) | Within 90 days from the index blood culture collection
  Number of participants with isolation of a new MDRO from recurrent positive blood cultures, or evidence of a worsened resistance profile compared to the index isolate
Incidence of Clostridioides difficile Infection (CDI) | Up to Day 28
  Number of participants with a laboratory-confirmed diagnosis of Clostridioides difficile infection
Incidence of Antibiotic-Related Adverse Events | Up to Day 28
  Number of participants experiencing adverse events (AE) judged by the investigator to be related to the antibiotic therapy (e.g., allergic reactions, renal toxicity)

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Cento, MD, PhD, Principal Investigator — Humanitas University
Locations (1):
- Microbiology and Virology - IRCCS Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Peled JU, Gomes ALC, Devlin SM, Littmann ER, Taur Y, Sung AD, Weber D, Hashimoto D, Slingerland AE, Slingerland JB, Maloy M, Clurman AG, Stein-Thoeringer CK, Markey KA, Docampo MD, Burgos da Silva M, Khan N, Gessner A, Messina JA, Romero K, Lew MV, Bush A, Bohannon L, Brereton DG, Fontana E, Amoretti LA, Wright RJ, Armijo GK, Shono Y, Sanchez-Escamilla M, Castillo Flores N, Alarcon Tomas A, Lin RJ, Yanez San Segundo L, Shah GL, Cho C, Scordo M, Politikos I, Hayasaka K, Hasegawa Y, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Jenq RR, Teshima T, Chao NJ, Holler E, Xavier JB, Pamer EG, van den Brink MRM. Microbiota as Predictor of Mortality in Allogeneic Hematopoietic-Cell Transplantation. N Engl J Med. 2020 Feb 27;382(9):822-834. doi: 10.1056/NEJMoa1900623. PMID 32101664
- [Background] Taur Y, Coyte K, Schluter J, Robilotti E, Figueroa C, Gjonbalaj M, Littmann ER, Ling L, Miller L, Gyaltshen Y, Fontana E, Morjaria S, Gyurkocza B, Perales MA, Castro-Malaspina H, Tamari R, Ponce D, Koehne G, Barker J, Jakubowski A, Papadopoulos E, Dahi P, Sauter C, Shaffer B, Young JW, Peled J, Meagher RC, Jenq RR, van den Brink MRM, Giralt SA, Pamer EG, Xavier JB. Reconstitution of the gut microbiota of antibiotic-treated patients by autologous fecal microbiota transplant. Sci Transl Med. 2018 Sep 26;10(460):eaap9489. doi: 10.1126/scitranslmed.aap9489. PMID 30257956
- [Background] von Dach E, Albrich WC, Brunel AS, Prendki V, Cuvelier C, Flury D, Gayet-Ageron A, Huttner B, Kohler P, Lemmenmeier E, McCallin S, Rossel A, Harbarth S, Kaiser L, Bochud PY, Huttner A. Effect of C-Reactive Protein-Guided Antibiotic Treatment Duration, 7-Day Treatment, or 14-Day Treatment on 30-Day Clinical Failure Rate in Patients With Uncomplicated Gram-Negative Bacteremia: A Randomized Clinical Trial. JAMA. 2020 Jun 2;323(21):2160-2169. doi: 10.1001/jama.2020.6348. PMID 32484534
- [Background] Giannella M, Pascale R, Toschi A, Ferraro G, Graziano E, Furii F, Bartoletti M, Tedeschi S, Ambretti S, Lewis RE, Viale P. Treatment duration for Escherichia coli bloodstream infection and outcomes: retrospective single-centre study. Clin Microbiol Infect. 2018 Oct;24(10):1077-1083. doi: 10.1016/j.cmi.2018.01.013. Epub 2018 Jan 31. PMID 29371138
- [Background] Yahav D, Franceschini E, Koppel F, Turjeman A, Babich T, Bitterman R, Neuberger A, Ghanem-Zoubi N, Santoro A, Eliakim-Raz N, Pertzov B, Steinmetz T, Stern A, Dickstein Y, Maroun E, Zayyad H, Bishara J, Alon D, Edel Y, Goldberg E, Venturelli C, Mussini C, Leibovici L, Paul M; Bacteremia Duration Study Group. Seven Versus 14 Days of Antibiotic Therapy for Uncomplicated Gram-negative Bacteremia: A Noninferiority Randomized Controlled Trial. Clin Infect Dis. 2019 Sep 13;69(7):1091-1098. doi: 10.1093/cid/ciy1054. PMID 30535100
- [Background] Mermel LA, Allon M, Bouza E, Craven DE, Flynn P, O'Grady NP, Raad II, Rijnders BJ, Sherertz RJ, Warren DK. Clinical practice guidelines for the diagnosis and management of intravascular catheter-related infection: 2009 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jul 1;49(1):1-45. doi: 10.1086/599376. PMID 19489710
- [Background] Stern A, Carrara E, Bitterman R, Yahav D, Leibovici L, Paul M. Early discontinuation of antibiotics for febrile neutropenia versus continuation until neutropenia resolution in people with cancer. Cochrane Database Syst Rev. 2019 Jan 3;1(1):CD012184. doi: 10.1002/14651858.CD012184.pub2. PMID 30605229
- [Background] Van de Wyngaert Z, Berthon C, Debarri H, Bories C, Bonnet S, Nudel M, Carpentier B, Legrand C, Barbieux S, Chauvet P, Simonnet A, Willaume A, Bossard JB, Renaud L, Wattebled KJ, Escure G, Branche N, Arib I, Titecat M, Quesnel B, Alfandari S. Discontinuation of antimicrobial therapy in adult neutropenic haematology patients: A prospective cohort. Int J Antimicrob Agents. 2019 Jun;53(6):781-788. doi: 10.1016/j.ijantimicag.2019.02.020. Epub 2019 Mar 2. PMID 30831232
- [Background] Aguilar-Guisado M, Espigado I, Martin-Pena A, Gudiol C, Royo-Cebrecos C, Falantes J, Vazquez-Lopez L, Montero MI, Rosso-Fernandez C, de la Luz Martino M, Parody R, Gonzalez-Campos J, Garzon-Lopez S, Calderon-Cabrera C, Barba P, Rodriguez N, Rovira M, Montero-Mateos E, Carratala J, Perez-Simon JA, Cisneros JM. Optimisation of empirical antimicrobial therapy in patients with haematological malignancies and febrile neutropenia (How Long study): an open-label, randomised, controlled phase 4 trial. Lancet Haematol. 2017 Dec;4(12):e573-e583. doi: 10.1016/S2352-3026(17)30211-9. Epub 2017 Nov 15. PMID 29153975
- [Background] Robilotti E, Holubar M, Seo SK, Deresinski S. Feasibility and applicability of antimicrobial stewardship in immunocompromised patients. Curr Opin Infect Dis. 2017 Aug;30(4):346-353. doi: 10.1097/QCO.0000000000000380. PMID 28542093
- [Background] Trecarichi EM, Pagano L, Martino B, Candoni A, Di Blasi R, Nadali G, Fianchi L, Delia M, Sica S, Perriello V, Busca A, Aversa F, Fanci R, Melillo L, Lessi F, Del Principe MI, Cattaneo C, Tumbarello M; HaematologicMalignancies Associated Bloodstream Infections Surveillance (HEMABIS) registry - Sorveglianza Epidemiologica Infezioni Funginein Emopatie Maligne(SEIFEM) group, Italy. Bloodstream infections caused by Klebsiella pneumoniae in onco-hematological patients: clinical impact of carbapenem resistance in a multicentre prospective survey. Am J Hematol. 2016 Nov;91(11):1076-1081. doi: 10.1002/ajh.24489. Epub 2016 Jul 29. PMID 27428072
- [Background] Gustinetti G, Mikulska M. Bloodstream infections in neutropenic cancer patients: A practical update. Virulence. 2016 Apr 2;7(3):280-97. doi: 10.1080/21505594.2016.1156821. PMID 27002635
- [Background] Mikulska M, Del Bono V, Bruzzi P, Raiola AM, Gualandi F, Van Lint MT, Bacigalupo A, Viscoli C. Mortality after bloodstream infections in allogeneic haematopoietic stem cell transplant (HSCT) recipients. Infection. 2012 Jun;40(3):271-8. doi: 10.1007/s15010-011-0229-y. Epub 2011 Dec 21. PMID 22187340
- [Background] Girmenia C, Bertaina A, Piciocchi A, Perruccio K, Algarotti A, Busca A, Cattaneo C, Raiola AM, Guidi S, Iori AP, Candoni A, Irrera G, Milone G, Marcacci G, Scime R, Musso M, Cudillo L, Sica S, Castagna L, Corradini P, Marchesi F, Pastore D, Alessandrino EP, Annaloro C, Ciceri F, Santarone S, Nassi L, Farina C, Viscoli C, Rossolini GM, Bonifazi F, Rambaldi A; Gruppo Italiano Trapianto di Midollo Osseo (GITMO) and Associazione Microbiologi Clinici Italiani (AMCLI). Incidence, Risk Factors and Outcome of Pre-engraftment Gram-Negative Bacteremia After Allogeneic and Autologous Hematopoietic Stem Cell Transplantation: An Italian Prospective Multicenter Survey. Clin Infect Dis. 2017 Nov 13;65(11):1884-1896. doi: 10.1093/cid/cix690. PMID 29020286
- [Background] Liu CY, Lai YC, Huang LJ, Yang YW, Chen TL, Hsiao LT, Liu JH, Gau JP, Chen PM, Tzeng CH, Chiou TJ. Impact of bloodstream infections on outcome and the influence of prophylactic oral antibiotic regimens in allogeneic hematopoietic SCT recipients. Bone Marrow Transplant. 2011 Sep;46(9):1231-9. doi: 10.1038/bmt.2010.286. Epub 2010 Nov 29. PMID 21113186
- [Background] Klastersky J. Management of fever in neutropenic patients with different risks of complications. Clin Infect Dis. 2004 Jul 15;39 Suppl 1:S32-7. doi: 10.1086/383050. PMID 15250018
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Zimmer AJ, Freifeld AG. Optimal Management of Neutropenic Fever in Patients With Cancer. J Oncol Pract. 2019 Jan;15(1):19-24. doi: 10.1200/JOP.18.00269. PMID 30629902